CLINICAL TRIAL: NCT06841393
Title: Knowledge and Exploratory Study to Better Understand Face Acne Pathophysiology and Acne Lesion Severity by Multi-omic Approaches, Biometrological Analysis and Consumer Needs
Brief Title: Assessment of Biological, Biometrological Parameters and Consumer Needs in Adult Subjects with Acne
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INTERACNE
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Acne; Healthy
MeSH Terms: conditions — Acne Vulgaris | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control subject group (Other)
  Interventions: Other: Biometrological measurements; Other: Biological sampling
- Subject group with mild to moderate acne on the face (Other)
  Interventions: Other: Biometrological measurements; Other: Biological sampling; Other: Clinical assessments; Other: Questionnaire

INTERVENTIONS:
Other: Biometrological measurements — Measurements will be taken from the face:
  * For acne group: inflammatory lesional area and non-lesional area
  * For control group: non-lesional area
Other: Biological sampling — Samples will be taken from the face:
  * For acne group: inflammatory lesional area, non-lesional area and retentional area
  * For control group: non-lesional area
Other: Clinical assessments — Only for acne group: acne scores will be evaluated on the face by the investigator
  Arms: Subject group with mild to moderate acne on the face
Other: Questionnaire — Only for acne group: consumers' perception
  Arms: Subject group with mild to moderate acne on the face

SUMMARY:
Acne vulgaris (acne) is a chronic inflammatory pathology of the pilosebaceous unit. Its prevalence is about 85% of teenagers and is constantly increasing in adults, especially women. Acne is a multifactorial disease involving abnormalities in follicular keratinization, sebum production, skin microbiota and inflammation.

The early stage of acne is characterized by the presence of primary retentional lesions: the open comedones (or blackheads) and closed comedones (or whitehead). These retentional lesions can progress to highly inflammatory lesions: superficial inflammatory lesions (papules and pustules) and in some cases in deep inflammatory lesions (nodules). Finally, acne lesions can lead to the development of superficial post inflammatory erythema or hyperpigmentation, resulting in emotional distress and a poorer quality of life.

Currently, a better understanding of the switch from healthy to acne-prone skin, but also of the transition from retentional lesions to more severe inflammatory lesions, seems essential to propose adapted and specific treatments.

The aim of this study is to better understand acne pathophysiology of the face by a multi-omic approaches, biometrological analysis and consumer needs collection to bring information, in the same study on the local ecosystem of non-lesional areas, retentional lesional areas and inflammatory lesional areas of adult acne prone skin, compared to acne free face.

ELIGIBILITY:
Inlcusion criteria:

Criteria related to the population:

* Subject aged between 18 and 30 years included
* For women of childbearing potential: use of an effective method of contraception, as assessed by the investigator, introduced and unchanged for at least 3 months before inclusion in the study

Criteria related to diseases:

Specific for acne group:

• Subject with acne lesions on the face, with a Global Acne Evaluation (GEA) score evaluated on the face of 2 (mild) or 3 (moderate) assessed by the investigator on a 5-point scale (0, 1, 2, 3, 4, 5 with 0 = clear - no lesions and 5 = very severe)

Non-inclusion criteria:

Criteria related to the population:

* For women of childbearing potential: pregnant or breastfeeding
* Subject having received on face artificial UV exposure, excessive or prolonged exposure to natural sunlight within 4 weeks before the inclusion visit
* Subject with facial hair liable to interfere with the study assessments

Criteria related to the disease:

* Clinical signs of hormone dysfunction or hyperandrogenism
* Severe form of acne (acne conglobata, acne fulminans or nodulocystic acne) or acneiform eruptions, in the investigator's opinion
* Sunburn on the face due to excessive UV exposure

Criteria related to skin condition:

• Subject having any other dermatologic condition than acne, or characteristics (like tattoo) on the face liable to interfere with the study assessments

Specific for control group:

* Subject with significant acne lesions according to investigator assessment
* Subject having any inflammatory face dermatosis

Criteria related to treatments and/or products:

* Any surgery, chemical or physical treatment on the face in the 12 months before the inclusion visit
* Systemic isotretinoin treatment taken in the 6 months prior before the inclusion visit
* Systemic acne treatment taken in the 3 months before the inclusion visit
* Probiotics taken orally in the month before the inclusion visit
* Topical acne treatment applied to the face in the month before the inclusion visit
* Topical or Systemic Non-Steroidal Anti-Inflammatory (NSAI), corticosteroids, taken or applied to the face in the 2 weeks before the inclusion visit
* Skincare product for acne liable to interfere with the study according to investigator's assessment applied to the face in the 2 weeks before the inclusion visit

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Cutaneous pH measurement | baseline (Visit 1- Day 1)
  by pH - pHmeter
Sebum quantification | baseline (Visit 1- Day 1)
  by Lipidic Index (LI) - Sebumeter®
Cutaneous barrier integrity | baseline (Visit 1- Day 1)
  by Trans-Epidermal Water Loss (TEWL) - Aquaflux®
Epigenetic analysis by sampling method (urine) | baseline (Visit 1- Day 1)
Microbiota profile by sampling method (swabs) | baseline (Visit 1- Day 1)
  By non-targeting metagenomics
Microbiota profile by sampling method (extracted comedones) | baseline (Visit 1- Day 1)
  for acne group only
Metabolomic profile by sampling method (swabs) | baseline (Visit 1- Day 1)
  By metabolomic analysis
Metabolomic profile by sampling method (extracted comedones) | baseline (Visit 1- Day 1)
  for acne group only
Lipidomic profile by mass spectroscopy (in-vivo measurements) | baseline (Visit 1- Day 1)
  Each characteristic peak corresponding to specific lipid will be quantified by its mass intensity
Lipidomic profile by sampling method (scotch) | baseline (Visit 1- Day 1)
  By lipidomic analysis
Lipidomic profile by sampling method (extracted comedones) | baseline (Visit 1- Day 1)
  for acne group only
Acne severity on the face | baseline (Visit 1- Day 1)
  using Global Acne Evaluation (GEA) scale on a 6-point scale (0, 1, 2, 3, 4, 5 with 0 = clear - no lesions and 5 = very severe) in acne group only
Lesions quantification | baseline (Visit 1- Day 1)
  by the number of inflammatory lesions (papules and/or pustules) in acne group
Consumers' perception | baseline (Visit 1- Day 1)
  by a questionnaire about acne skin, skincare routine, needs and expectations in terms of facial care in acne group

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Research Center, Toulouse, France